CLINICAL TRIAL: NCT01181544
Title: Heparin Dose Reduction During Hemodialysis With the Gambro Revaclear and Revaclear MAX Hemodialyzers: Pilot Study I and II
Brief Title: A Pilot Study of a Heparin Dosing Algorithm for Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: University of Louisville (Other); Gambro Renal Products, Inc. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gambro PI 2012
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis
Keywords: Anticoagulation; Heparin; Hemodialysis; Dialysis; Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heparin dose titration (Experimental)
  Interventions: Procedure: Heparin dose titration

INTERVENTIONS:
Procedure: Heparin dose titration — Patients will begin the study using their currently prescribed heparin doses - both bolus and constant infusion - for three treatments to establish a baseline and provide information on inter-treatment variability in dialyzer clotting. Subsequently, the bolus and infusion rates will be titrated either upward or downward based on the Robbins-Monro process and an evaluation of dialyzer clotting during the preceding treatment. Heparin doses will be adjusted for a total of 30 dialyses.

SUMMARY:
During hemodialysis treatments, patients receive heparin to prevent clotting. The purpose of this pilot study is to determine if the amount of heparin administered during a patient's hemodialysis can be individualized using an equation for heparin dose adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Stable hemodialysis prescription prior to study enrollment
* Dialyzing through a native fistula or Gore-Tex graft
* Blood access must be able to provide a blood flow rate of 400 ml/min

Exclusion Criteria:

* Non-compliance with dialysis
* Hematocrit less than 28%
* Active Infection
* Diagnosis of Heparin-Induced Thrombocytopenia (HIT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in dialyzer blood compartment volume when the heparin dose is adjusted using a Robbins-Monro algorithm | up to 8 weeks
  The objective is to titrate each patient's heparin dose to the level that achieves adequate anticoagulation for that patient as assessed by the change in blood compartment volume of the dialyzer from pre- to post-dialysis. The strategy that will be used is the Robbins-Monro stochastic approximation algorithm.

SECONDARY OUTCOMES:
Evaluation of dialyzer performance and visual assessment of clotting in the fiber bundle and the arterial and venous headers | up to 8 weeks
  Visual assessment of the dialyzer,measurement of ionic dialysance and ionic Kt/V.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Ward, Ph.D., Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Background] Farrell PC, Ward RA, Schindhelm K, Gotch F. Precise anticoagulation for routine hemodialysis. J Lab Clin Med. 1978 Aug;92(2):164-76. PMID 681809
- [Background] Smith BP, Ward RA, Brier ME. Prediction of anticoagulation during hemodialysis by population kinetics and an artificial neural network. Artif Organs. 1998 Sep;22(9):731-9. doi: 10.1046/j.1525-1594.1998.06101.x. PMID 9754457
- [Background] Robbins H, Monro S. A stochastic approximation method. Ann Math Stat 22:400-407, 1951.
- [Background] Association for the Advancement of Medical Instrumentation: Reuse of Hemodialyzers (ANSI/AAMI RD47:2003). Association for the Advancement of Medical Instrumentation, Arlington, VA, 2003.